CLINICAL TRIAL: NCT02944799
Title: Alendronate Treatment of Osteoporosis in Rheumatoid Arthritis - Indication and Duration: A Randomized, Double-blind, Placebocontrolled Study to Evaluate the Effects of Discontinuation of Alendronate in Patients With Both Rheumatoid Arthritis and Low Bone Mass
Brief Title: Alendronate Treatment of Osteoporosis in Rheumatoid Arthritis
Acronym: ALOSTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-003638-28
Record Dates: First submitted 2016-06-27; First posted 2016-10-26 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis; Osteoporosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis | interventions — Alendronate; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Active Comparator): Continues treatment with alendronate, 70mgs oral tablet once every week
  Interventions: Drug: Alendronate; Drug: Calcium; Drug: Vitamin D
- Placebo (Placebo Comparator): Placebo tablets, one every week
  Interventions: Drug: Placebo; Drug: Calcium; Drug: Vitamin D

INTERVENTIONS:
Drug: Placebo — Discontinuation of alendronate treatment
  Arms: Placebo
Drug: Alendronate
  Arms: Alendronate
Drug: Calcium — Daily dietary supplement of 800mg calcium
Drug: Vitamin D — Daily dietary supplement of 38 micrograms vitamin D

SUMMARY:
A randomized, double-blind, placebo-controlled trial including 160 consecutive patients who have been diagnosed with both rheumatoid arthritis (RA) and low bone mass and have been treated with alendronate (ALN) for five years or more. Patients will be randomized to discontinuation or continuation of alendronate. Outcomes are measured using dual energy absorptiometry (DXA), High Resolution peripheral Quantitative Computer Tomography (HR-pQCT) and biochemical markers of bone metabolism and inflammation after 6 months, 1 and 2 years.

DETAILED DESCRIPTION:
Primary objectives:

* to assess the effect of discontinuation of alendronate (ALN) on C-terminal telopeptide crosslinks (CTX) and Type 1 procollagen amino-terminal-propeptide (P1NP) after 6 months
* to assess the effect of discontinuation of ALN on bone mineral density (BMD) on DXA scans at 2 years

Secondary objectives:

* to assess the effect of discontinuation of ALN on vBMD on HRpQCT scans at 2 years
* to assess the effect of discontinuation of ALN on biochemical markers of bone metabolism after 6 and 24 months
* to evaluate and compare the changes in vBMD in cancellous and cortical bone respectively, after discontinuation of ALN
* to evaluate the correlation between RA activity measured by DAS28-CRP and bone metabolism

Interventions:

Participants will be randomized to one of two groups:

* Group 1 (Alendronate group, N=80): alendronate 70mg/weekly, calcium 800 mg/day and vitamin D 38 µg/day
* Group 2 (Placebo group, N=80): alendronate-placebo, calcium 800 mg/day and vitamin D 38 µg/day

Concomitant treatment of RA:

Patients included in this trial will be treated according to the national Danish guidelines for treatment of RA

Assignment of intervention:

The Hospital Pharmacy in Aarhus will carry out the randomization. Using the web-based programme randomization.com a list of distribution is produced. The randomization will be stratified according to which type of treatment the patients receives for RA. All patients receiving traditional DMARDs such as methotrexate, sulfasalazine, hydroxychloroquine, leflunomide or a combination hereof will be allocated to grop A. All patients receiving any kind of biological treatment (bDMARDs) e.g. infliximab will be allocated to group B. When requesting randomization from the hospital pharmacy, the investigator will note if the patient is group A or B. Both group A and B will undergo randomization 1:1 in the ALN and placebo groups, using block randomization in blocks of 6.

Participant timeline:

Patients will be seen at a screening visit, at baseline and after 3, 6, 12, and 24 months

Procedures at screening: informed consent procedures, full medical history, full physical examination, 12- lead EKG, screening blood samples, DXA scan

Procedures at all other visits: focused physical exam of joints and back, measurement of blood pressure, pulse and temperature, calculation of DAS28-CRP and HAQ scores, screening for adverse events, routine and project blood samples.

At baseline visit: HRpQCT scan and Xrays of hands and feet

At visit 12 months: DXA and HRpQCT scans

At visit 24 months: DXA and HRpQCT scans, xrays of hands and feet

Clinical laboratory tests:

* routine analyses include: alkaline phosphatase, creatinine, alanine aminotransferase (ALT), platelet count, Hemoglobin, white blood cells, absolute neutrophil count, absolute lymphocyte count, CRP (total 8ml)
* screening analyses: routine analysis as well as s-FSH and/or HCG (women only), calcium, PTH, vitamin-D status, TSH (total 16 ml)
* primary project analyses include: CTX and P1NP (total 4 ml)
* secondary project analysis include: bone specific alkaline phosphatase, RANK-L, sclerostin, tumor necrosis factor, osteoprotegrin, P1NP, osteocalcin, IL-6, IL-17 (total 8 ml)
* extra blood bank sample - 3ml serum, 2 ml plasma and full blood for storage and later analysis

DXA scan:

Study participants will be scanned using a Hologic discovery machine.To ensure comparative results, the same machine will be used for each participant at each scan. Lumbar spine anterior-posterior and left hip pictures are recorded following local guidelines.

HR-pQCT scan:

Bone structure will be measured at metacarpals 2-4 and proximal radius using the model XTREME CT-I SCANCO MEDICAL AG; SCHWEIZ. A 2,7 cm long area over the right hand second and third metacarpophalangeal joint is scanned. After this a 0,9 cm long part of the distal radius is scanned The 3D dataset will be analyzed and number and volume of erosions calculated. Volumetric BMD is calculated for both cortical and trabecular bone, trabecular number and separation according to the built-in software.

X-rays of hands and feet:

Standardized X-rays of the hands/forearms and upper feet in separate AP (dorsopalmar) projections of each hand and wrist and dorsoplantar projections of the feet Images of the hands will be centered around the 2nd and 3rd MCPjoints The foot must not be tilted in the case of suboptimal projections of the MTP-joints. All images will be scored centrally according to the Sharp-van der Heide score system.

DAS28-CRP:

A clinical activity score for arthritis activity is calculated by means of

* number of tender and swollen joint scores including the following twenty eight joints: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees.
* crp-measurement
* general health assessment by the doctor using a VAS-scale A number between 0 and 10 is calculated. Values <2,6 are considered in remission, values >2,6 are considered as evidence of disease activity

Harms:

The dose of radiation is estimated to 0,07mSievert, as each HR-pQCT scan contributes with 0,012mS, each DXAscan 0,01mS and each Xray status of hands and feet 0,008mS. The average annual background radiation exposure in Denmark is 3mSievert. Thus the participants will receive an increased radiation dose corresponding to 9 days of background radiation.

The HR-pQCT-scans require fixation of the hand for 8 and 3 minutes respectively, which might cause slight discomfort.

Safety measures:

All routine biochemical markers (visit 1-5) will be analyzed and evaluated promptly. An increase in alkaline phosphatase of more than 100% will lead to the participant being called in for an extra visit for further evaluation of the cause. The patient will be withdrawn from the study if there is suspicion of accelerated bone loss.

All fractures will be recorded and in the case of low-energy fracture the patient will be withdrawn from the study.

The 12 month DXA scans will be reviewed and a BMD decrease of more than 5% will lead to exclusion from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients (> 18 years) with rheumatoid arthritis according to the ACR(1987 or 2010)/EULAR (2010) classification criteria (12)
* treated with alendronate for five years or more
* current T-score on DXA better than or equal to -2,5 (femoral) and -3,0 (vertebral)
* receiving treatment on an outpatient basis
* negative pregnancy test (serum HCG) prior to trial start and the use of contraception throughout the study period and for 1 month after conclusion of the study period for women of childbearing potential. Plasma T1/2 of ALN is less than 2 hours. The forms of contraception include: intrauterine device (IUD) and hormonal anticontraceptives (contraceptive pill, implant, patch or injection or vaginal ring). Sterile and non-fertile participants do not have to use contraception. Sterile or non-fertile is defined as having undergone surgical sterilization (vasectomy / bilateral tubectomy, hysterectomy and bilateral oophorectomy) or post-menopausal status, defined as absence of menstrual period for at least 12 months prior to enrollment. Postmenopause will be confirmed by measurement of s-FSH prior to enrollment.
* ability and willingness to give written informed consent and to meet the requirements of the trial protocol.

Exclusion Criteria:

* history of hip fracture due to osteoporosis
* history of vertebral fracture of more than one vertebrae or other fragility fractures within the last three years (fingers and toes not included)
* osteonecrosis of the jaw.
* history of or ongoing systemic GC treatment within the last 6 months (intraarticular injections are approved)
* known allergy toward any components of the study medicine
* prior or ongoing treatment with other antiosteoporosis drugs such as hormone replacement therapy or teriparatide
* active malignant disease
* metabolic bone disease other than osteoporosis
* hypo- or hyperthyroidism
* hypocalcaemia
* impaired renal function (eGFR <35ml/min)
* known disease of the esophagus that might impair the ability to swallow the tablets such as achalasia, dysphagia or strictures
* history of upper gastrointestinal disease within 1 year prior to enrollment such as peptic ulcer, upper GI bleeding, gastritis, duodenitis or surgical procedures to the upper GI-tract
* allergy towards any of the substances in the study medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Change from baseline to 24 months
C-terminal telopeptide crosslinks (CTX) | Change from baseline to 6 months
  serological marker of bone metabolism
Type 1 procollagen amino-terminal-propeptide (P1NP) | Change from baseline to 6 months
  serological marker of bone metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hauge, MD, PhD, Principal Investigator — University of Aarhus
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Hjørring Hospital, Hjørring
  - Odense University Hospital, Odense
  - Silkeborg Regional Hospital, Silkeborg
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided